CLINICAL TRIAL: NCT00557115
Title: Early Pulmonary Rehabilitation (PR) Following Hospitalisation For Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Early Pulmonary Rehabilitation Following Acute COPD Exacerbation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: British Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/Q0703/093; BLF PO4/8
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2007-11

CONDITIONS: COPD
Keywords: Quality of life; Quadriceps; Muscle; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Usual Care (UC): usual follow up care post acute COPD exacerbation
- EPR (Experimental): Early pulmonary rehabilitation (EPR): pulmonary rehabilitation commenced within 1-week of hospital discharge from an acute COPD exacerbation
  Interventions: Other: Early pulmonary rehabilitation (EPR)

INTERVENTIONS:
Other: Early pulmonary rehabilitation (EPR) — Multidisciplinary exercise programme in the format of standard pulmonary rehabilitation. Consists of 2 supervised exercise and educations sessions per week for up to 16 sessions within 3-months. Participants are encouraged to keep an exercise diary at perform at least one exercise session at home unsupervised.
  Arms: EPR

SUMMARY:
The principal aim of the study is to evaluate whether attendance at an exercise training and education programme (known as pulmonary rehabilitation) shortly following hospital discharge can lead to a reduction in exacerbations and improvement in exercise capacity and quality of life in patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Background:

Chronic obstructive pulmonary disease (COPD), also sometimes known as chronic asthma, bronchitis or emphysema, is an important health problem. Many people with COPD are admitted into hospital with a worsening of their symptoms, known as an exacerbation. Hospitalisations for acute exacerbations of chronic obstructive pulmonary disease (COPD) are a massive burden to the NHS. Over the past decade, these hospitalizations have increased by 50%, and annual hospital costs for COPD in the UK amount to more than £587 million. After being discharged, some people fail to cope very well due to a variety of reasons. A prolonged stay in hospital may lead to muscle weakness, particularly of the leg muscles [1], a loss of confidence in performing everyday activities, and increased anxiety [2]. A high proportion of these patients are re-admitted to hospital following discharge. The aim of the study is to assess whether attendance at an exercise training and education programme shortly following discharge can firstly, improve exercise capacity and quality of life, and secondly, reduce the use of health resources and costs to the NHS.

It is known that an exercise training and education programme known as Pulmonary Rehabilitation is beneficial to stable patients with COPD by reducing breathlessness, increasing exercise capacity and improving quality of life. We have recently performed a pilot study that has shown that early Pulmonary Rehabilitation has considerable short-term benefits in patients with COPD who have been recently discharged following a hospital admission for worsening of their symptoms [3]. We hypothesise that these benefits are long-lasting, and may reduce use of healthcare resources and costs to the NHS.

References:

1. Spruit, M.A., et al., Muscle force during an acute exacerbation in hospitalised patients with COPD and its relationship with CXCL8 and IGF-I. Thorax, 2003. 58(9): p. 752-6.
2. Seemungal, T.A., et al., Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med, 1998. 157(5 Pt 1): p. 1418-22.
3. Man, W.D., et al., Community pulmonary rehabilitation after hospitalisation for acute exacerbations of chronic obstructive pulmonary disease: randomised controlled study. BMJ, 2004. 329(7476): p. 1209.

Description of Study:

Based on the results of our pilot study [1], we hypothesise that early pulmonary rehabilitation (EPR) leads to long term improvements in exercise capacity, quality of life, use & resulting costs of healthcare resources, peripheral muscle strength and daily activity levels. The null hypothesis is that EPR does not lead to a significant difference in outcome when compared to usual care (UC).

EXPERIMENTAL DESIGN AND METHODS: This is a prospective randomised controlled clinical trial of EPR vs. usual care.By using a control group, statistically significant differences in outcome can be attributed to EPR. No treatment considered to be part of routine care is being withheld from the UC group.

Patients: Patients studied will be those with an acute exacerbation of COPD deemed sufficiently unwell by the duty medical registrar to warrant hospital admission. Exclusion criteria will include significant co-morbidity that could limit exercise training, and attendance at a pulmonary rehabilitation programme in the preceding year. In-patient treatment will include standard therapy (nebulised bronchodilators, oxygen, non-invasive ventilation (if required), antibiotics and a 1-2 week course of oral prednisolone 30-40mg daily). On hospital discharge, patients will be allocated either to the early pulmonary rehabilitation (EPR) group (within 7 days of hospital discharge) or usual care (UC) i.e. routine outpatient and primary-care follow-up.

PROTOCOL: In the 48 hours before planned hospital discharge, the following measurements will be made in all patients:

1. Pulmonary function tests, including ear-lobe blood gases, spirometry, lung volumes, and transfer factor.
2. Anthropometric data, including height, weight, body mass index, lean body mass (as measured by bio-electrical impedance)
3. Field exercise capacity as measured by the incremental shuttle walk, a standard externally paced, incremental, maximal,corridor-walking test [2].
4. Disease-specific and generic health status, as measured by the Chronic Respiratory Diseases Questionnaire (CRDQ) [3],St George's Respiratory Questionnaire (SGRQ) [4]. Interviews will take place in the lung function department at King's College Hospital.
5. Cardiopulmonary exercise testing in a subset of voulnteers, with measurements of VO2, and VCO2 and lactic acid.
6. Non-volitional and volitional quadriceps strength: twitch quadriceps tension following supramaximal stimulation of femoral nerve and maximum isometric voluntary contraction. This is a painless supramaximal method of assessing quadriceps strength and fatigue [5] [6].
7. Endurance walking capacity (endurance shuttle walk)
8. Health resource usage (see later). The EuroQol (EQ-5D) instrument [7] will be used as the main measure of health-related quality-of-life in the economic evaluation.

The measurements made at baseline will be repeated at 3 and 12 months. Of note, as this study is a prospective longitudinal study, patients will be familiarised with the exercise tests in the days before discharge to minimise learning effect. Verbal encouragement during exercise testing will be standardised to avoid researcher effects. The assessor will be blinded to the subject's intervention. However owing to the nature of the intervention, it will not be possible to blind the subjects to their intervention.

RANDOMISATION: At discharge, patients will be allocated to either a hospital outpatient exercise rehabilitation programme, or usual care. Due to the numbers to be studied, allocation of treatments using the minimisation method will be used to ensure comparable groups. The following factors will be taken into account:

1. Age (above and below 70)
2. Gender (male/female)
3. Hospital Discharge incremental shuttle walk distance (more or less than 100 metres).
4. Length of Hospital Admission (more or less than 7 days)
5. FEV1 more or less than 30% predicted

INTERVENTION: Patients allocated to the EPR group will attend a pulmonary rehabilitation programme within 7 days of hospital discharge. This will consist of two sessions a week for 8 weeks, and will be supervised by a multi-disciplinary team consisting of physiotherapists, occupational therapists, nurses and dieticians as well as the clinical research fellow funded by the proposed grant. Each session consists of 60 minutes exercise, made up of aerobic walking and cycling exercise plus lower and upper limb strength and endurance exercise, and 1 hour of discussion focusing on psychosocial and lifestyle issues, with a particular emphasis on nutrition and domestic activity. The EPR group will be also be given an individualised home exercise programme, encouraging daily exercise. The UC group will receive usual outpatient and primary care follow-up.

HEALTH ECONOMICS: The EuroQol (EQ-5D) instrument will be used as the main measure of health-related quality-of-life in the economic evaluation [9]. It has been developed by a collaborative group of European researchers as a preference-based index, suitable for the calculation of QALYs. The EQ-5D is one of two instruments currently recommended for use in economic evaluations [8]. Information on patients' use of health services will be collected by a review of hospital notes, patient recall and a home diary issued to all study participants. The resources included will be: hospital admissions, inpatient days, ITU days, outpatient consultations, A&E attendances, and primary care surgery and home visits.

SAMPLE SIZE: Our preliminary pilot study was powered to detect a 50-metre difference in incremental shuttle walk at the 5% significance level with 90% power. Based on the health resource usage data collected from this pilot study, to detect a 50% reduction in hospital readmission rate at the 5% significance level with 80% power would require a minimum of 60 patients (30 in each group). We propose to study 80 patients in this study

References:

1. Man, W.D., et al., Community pulmonary rehabilitation after hospitalisation for acute exacerbations of chronic obstructive pulmonary disease: randomised controlled study. BMJ, 2004. 329(7476): p. 1209.
2. Singh, S.J., et al., Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax, 1992. 47(12): p. 1019-24.
3. Guyatt, G.H., et al., A measure of quality of life for clinical trials in chronic lung disease. Thorax, 1987. 42(10): p. 773-8.
4. Jones, P.W., et al., A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis, 1992. 145(6): p. 1321-7.
5. Man, W.D., et al., Non-volitional assessment of skeletal muscle strength in patients with chronic obstructive pulmonary disease. Thorax, 2003. 58(8): p. 665-9.
6. Polkey, M.I., et al., Quadriceps strength and fatigue assessed by magnetic stimulation of the femoral nerve in man. Muscle Nerve, 1996. 19(5): p. 549-55.
7. Brooks, R., EuroQol: the current state of play. Health Policy, 1996. 37(1): p. 53-72.
8. Brazier, J., M. Deverill, and C. Green, A review of the use of health status measures in economic evaluation. J Health Serv Res Policy, 1999. 4(3): p. 174-84.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to King's College Hospital with a clinical diagnosis of acute exacerbation of COPD. Patients with radiological and microbiological evidence of pneumonia with co-existing COPD will also be included.

Exclusion Criteria:

* Significant co-morbidity that could limit exercise training & testing: Patients unable to walk due to a comorbid neuromuscular or rheumatological condition; patients with severe sensory and cognitive impairment; patients with unstable angina or aortic valve disease in which exercise could be dangerous.
* Attendance at a pulmonary rehabilitation programme in the preceding year.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-04-15 (Actual); Study Completion 2008-04-16 (Actual)

PRIMARY OUTCOMES:
Non-outpatient COPD related hospital attendance (A+E attendance, inpatient admission or death) | 3-months

SECONDARY OUTCOMES:
Disease specific quality of life (CRDQ and SGRQ) | 3 months and 1-year
Maximal walking capacity (ISW)and endurance walking capacity (ESW) | 3-months and 1-year
Weight and fat free mass (electrical bioimpedance) | 3-months and 1-year
Quadriceps muscle strength (volitional and non-volitional) | 3-months and 1-year
Cost-effectiveness (Index derived from EQ-5D) | 3-months and 1-year

CONTACTS AND LOCATIONS:
Overall Officials: John Moxham, MD FRCP, Principal Investigator — King's College London
Locations (3):
- United Kingdom (3):
  - Basildon University Hospital, Basildon, Essex
  - St Thomas' Hospital, London
  - King's College Hospital, London

REFERENCES:
- [Derived] Seymour JM, Moore L, Jolley CJ, Ward K, Creasey J, Steier JS, Yung B, Man WD, Hart N, Polkey MI, Moxham J. Outpatient pulmonary rehabilitation following acute exacerbations of COPD. Thorax. 2010 May;65(5):423-8. doi: 10.1136/thx.2009.124164. PMID 20435864